CLINICAL TRIAL: NCT01458639
Title: A Comparison of Technegas® Ventilation-Perfusion SPECT and Xenon Ventilation-Perfusion Planar Imaging in Subjects Being Evaluated for Pulmonary Embolism
Brief Title: Compare Technegas Ventilation-Perfusion SPECT and Xenon Ventilation-Perfusion Planar Imaging for Pulmonary Embolism
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Decision to change trial design.
Sponsor: Cyclomedica Australia PTY Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: CYC-008
Record Dates: First submitted 2011-10-19; First posted 2011-10-25 (Estimated); Results first posted 2015-11-10 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-10

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary embolism; PE
MeSH Terms: conditions — Pulmonary Embolism | interventions — Technetium; Xenon-133

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Technegas (Experimental): Technegas V SPECT imaging with Technetium-99m (Tc-99m) labeled carbon particles; approximately 1.1 milliCuries of Technegas, compared with the results of Xenon-133 ventilation scan
  Interventions: Drug: Technegas V SPECT imaging
- Xenon-133 (Active Comparator): Xenon-133 ventilation Planar imaging compared with the results of the Technegas scan.
  Interventions: Drug: Xenon-133 Ventilation Planar imaging

INTERVENTIONS:
Drug: Technegas V SPECT imaging — Technegas V SPECT imaging and Technetium 99m MAA Perfusion imaging for the diagnosis pf pulmonary embolism.
  Other Names: Technetium-99m (Tc-99m) labeled carbon particles
  Arms: Technegas
Drug: Xenon-133 Ventilation Planar imaging — Xenon-133 Ventilation Planar imaging and Technetium 99m MAA Perfusion imaging for the diagnosis pf pulmonary embolism.
  Other Names: Xe-133
  Arms: Xenon-133

SUMMARY:
Phase 3 within-subject trial of Technegas V/Q SPECT and Tc-99m macro-aggregated albumin (MAA) imaging compared to Xenon-133 V/Q planar and Tc-99m macroaggregate of albumin (MAA) imaging for the diagnosis of Pulmonary Embolism (PE).

DETAILED DESCRIPTION:
This is a Phase 3 within-subject trial of Technegas Ventilation SPECT and Tc-99m MAA perfusion imaging compared to xenon (Xe-133) Ventilation Planar and Tc-99m MAA perfusion imaging for the diagnosis of PE. Diagnosis of PE provided by review of the subjects' documented clinical information after 30 days of follow-up. Primary assessments of efficacy will be based on an independent blind reads of the Technegas V/Q SPECT images by three different readers and the independent blind reads of Xe 133 V/Q planar images by three different readers.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be enrolled in Cohort 1 if they meet the following requirements:

1. Male or female, at least 18 years of age.
2. Suspected of having PE and be a candidate for Xe-133 V/Q imaging.
3. Willing and able to provide informed consent.
4. Stable and able to undergo Xe-133 planar imaging, Technegas SPECT imaging, and planar/SPECT perfusion imaging and complete follow-up procedures.
5. Willing and agree to complete study procedures, including follow-up safety assessments.
6. Using adequate birth control, if female and fertile.
7. If female, has a negative urine or serum pregnancy test.
8. Agrees to return for a 24-hour and 30 day follow-up safety assessment.

Subjects will be enrolled in Cohort 2 if they meet the above criteria AND subject is likely to have pulmonary embolism based on one or more of the following:

1. Wells Score of 7 or greater. Subjects with a Wells Score less than 7 may be enrolled in Cohort 2 if there is agreement between the investigator and the medical monitor that the subject is at high risk for PE.
2. An abnormal D-dimer test.
3. Positive Doppler ultrasound for DVT.
4. CTA is positive for PE within 24 hours of this imaging study.

Exclusion Criteria:

Subject

1. Has undergone imaging with Iodine-131 (I-131) within 30 days, Thallium-201 (Tl-201) or Indium-111 (In-111) within 10 days, Fluorine 18 (F-18) within 24 hours, or any other radiopharmaceutical not otherwise specified within 72 hours of this imaging study.
2. Has previously undergone an imaging study with a Tc-99m agent, within 48 hours of this imaging study.
3. Is a pregnant or lactating female.
4. Has received Technegas in the past.
5. Was previously enrolled in another investigational study or received an investigational drug within 30 days prior to dosing.
6. Is hemodynamically unstable.
7. Has received therapeutic dose of low molecular weight or unfractionated heparin within 24 hours prior to dosing or Tissue Plasminogen Activator (tPA) within 4 hours prior to dosing or has received treatment for PE between the time of a positive CTA, if performed, and Technegas V/Q SPECT imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward M Aten, MD, Study Director — Certus International, Inc.; Akash Sharma, MD, Principal Investigator — Washington University Mallinckrodt Institute of Radiology; David Leung, MD, PhD, Principal Investigator — Columbia University Medical Center, New York, NY
Locations (2):
- United States (2):
  - Barnes-Jewish Hospital, Washington University, St Louis, Missouri
  - Columbia University Medical Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was November 14, 2012 to June 11, 2014. Subjects were recruited from US medical centers that performed Xenon-133 ventilation scans to evaluate patients for pulmonary embolism (PE).
Pre-assignment Details: Subjects suspected of PE to have Xe-133 ventilation/Tc-99m macroaggregated albumin (MAA) perfusion (VQ) scan. Must have at least one within 72 hours before imaging: D-dimer, Doppler ultrasound for deep vein thrombosis (DVT) or computed tomography angiography (CTA) for PE. Not have therapeutic dose blood thinner for > than 72 hrs prior to imaging.
Groups:
- Overall Study: Xenon-133 Ventilation Planar imaging, followed by Technegas Ventilation SPECT imaging with Technetium-99m (Tc-99m) labeled carbon particles, followed by Technetium 99m (Tc-99m) MAA Perfusion imaging for the diagnosis of pulmonary embolism. Xe-133 V / Tc-99m MAA Q results compared to Technegas V / Tc-99m MAA Q results.
Period: Overall Study
Arm/Group | Overall Study
Started | 18
Completed | 12
Not Completed | 6
Not completed — Physician Decision | 4
Not completed — Equipment issue | 1
Not completed — Inability to obtain subject blood sample | 1

BASELINE CHARACTERISTICS:
Population: All subjects enrolled in the trial.
Arm/Group | Overall Study
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 6
Age, Continuous [Mean (Full Range); unit: years] | 59.5 [34 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of Technegas V/Q SPECT for the Diagnosis of PE
Description: Compared to the sensitivity of Xenon V/Q Planar imaging. "Truth" based on blinded reader's assessments of V/Q SPECT images compared with subject's final diagnosis resulting from clinical information at 30 days follow-up.
Time Frame: Prospective, 30 days follow-up
Population: Pulmonary embolism adjudication was to be determined by an Independent Adjudication Committee for primary and secondary outcome data and blinded readings of Xe-133 and Technegas Ventilation and Tc-99m MAA Perfusion images were required for primary outcome data. Due to trial termination PE adjudication and blinded readings of images were not done.
Arm/Group | Overall Study
Number analyzed (Participants) | 0

2. Primary Outcome: Specificity of Technegas V/Q SPECT for the Diagnosis of PE.
Description: Compared to the specificity of Xenon V/Q Planar imaging. "Truth" based on blinded reader's assessments of V/Q SPECT images compared with subject's final diagnosis resulting from clinical information at 30 days follow-up.
Time Frame: Prospective, 30 days follow-up
Population: as for outcome 1
Arm/Group | Overall Study
Number analyzed (Participants) | 0

3. Secondary Outcome: Accuracy of Technegas V/Q SPECT and Xenon V/Q Planar Imaging for Diagnosis of PE
Description: Accuracy of V/Q imaging for diagnosis of PE is determined by the results of blind-read assessment of images compared with truth using a subject's final clinical diagnosis following 30-day follow-up of occurence of PE or death, whichever occurs first.
Time Frame: prospective, 30 days follow-up.
Population: PE adjudication for final clinical diagnosis was to be determined by an Independent Adjudication Committee and blinded readings of Xe-133 and Technegas Ventilation and Tc-99m MAA Perfusion images were required for primary and secondary outcome data. Due to trial termination PE adjudication and blinded readings of images were not done.
Arm/Group | Overall Study
Number analyzed (Participants) | 0

4. Secondary Outcome: Positive Predictive Value (PPV) of Imaging for Diagnosis of PE
Description: PPV of V/Q imaging for diagnosis of PE is determined by the results of blind-read assessment of images compared with truth using a subject's final clinical diagnosis following 30-day follow-up of occurence of PE or death, whichever occurs first.
Time Frame: Prospective, 30 days follow-up
Population: as for outcome 3
Arm/Group | Overall Study
Number analyzed (Participants) | 0

5. Secondary Outcome: Negative Predictive Value (NPV) of Imaging for Diagnosis of PE
Description: NPV of V/Q imaging for diagnosis of PE is determined by the results of blind-read assessment of images compared with truth using a subject's final clinical diagnosis following 30-day follow-up of occurence of PE or death, whichever occurs first.
Time Frame: Prospective, 30 days follow-up
Population: as for outcome 3
Arm/Group | Overall Study
Number analyzed (Participants) | 0

6. Secondary Outcome: Likelihood Ratio for Diagnosis of PE
Description: Likelihood ratios of V/Q imaging for diagnosis of PE is determined by the results of blind-read assessment of images compared with truth using a subject's final clinical diagnosis following 30-day follow-up of occurence of PE or death, whichever occurs first.
Time Frame: Prospective, 30 days follow-up
Population: as for outcome 3
Arm/Group | Overall Study
Number analyzed (Participants) | 0

7. Secondary Outcome: Safety of Technegas in Patients With Possible PE
Description: Safety will be assessed by the incidence of treatment emergence adverse events and changes in clinical laboratory measurements, blood pressure, oxygen saturation, physical examination and pulmonary examination before and after treatment.
Time Frame: Prospective, from enrollment through 30 days follow-up
Population: All subjects who received Technegas and completed safety follow-up procedures.
Measure: Number; unit: participants
Arm/Group | Overall Study
Number analyzed (Participants) | 12
participants
  Serious adverse events | 0
  Other (not including serious) adverse events | 1

ADVERSE EVENTS:
Time Frame: 24 (+/- 4) hours post Technegas ventilation/perfusion (V/Q) scan.
Description: Safety assessment was performed from the start of the Xe-133 ventilation scan, followed by the Technegas ventilation scan, followed by the Tc-99m MAA scan until 24 (+/- 4) hours after the Technegas ventilation scan.
Arm/Group | Overall Study
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Study (N=12)
Systolic blood pressure increase (Investigations) | 1 (1) — 24 min. post Technegas administration, subject had increase in systolic blood pressure (SBP) from 103 to 140 mmHg (increase of 37) meeting protocol definition SBP increase > 35 mmHg being clinically significant. Resolved spontaneously in 2 min.

LIMITATIONS AND CAVEATS:
PE adjudication by Independent Committee for final clinical diagnosis and blinded readings of Xe-133 and Technegas Ventilation and Tc-99m MAA Perfusion images were not performed due to early trial termination. No efficacy data available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No